CLINICAL TRIAL: NCT03731182
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Comparator Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 in Children With Sickle Cell Disease (PNEU-SICKLE)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 in Children With Sickle Cell Disease (V114-023/PNEU-SICKLE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-023; V114-023 (Other: Merck Protocol Number); 2018-001152-35 (EudraCT Number)
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V114 on Day 1.
  Interventions: Biological: V114
- Prevnar 13™ (Active Comparator): Participants will receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1.
  Interventions: Biological: Prevnar 13™

INTERVENTIONS:
Biological: V114 — V114 pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, 33F (2 mcg each), and serotype 6B (4 mcg) in each 0.5 mL dose
  Arms: V114
Biological: Prevnar 13™ — Prevnar 13™ pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg) and 6B (4.4 mcg) in each 0.5 ml dose
  Arms: Prevnar 13™

SUMMARY:
This study is designed to describe the safety, tolerability, and immunogenicity of V114 in children with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of sickle cell disease in their medical record
* Female participants: not pregnant or breastfeeding, and at least 1 of the following conditions apply:

  1) not a woman of childbearing potential (WOCBP) as defined in the protocol, or 2) a WOCBP who agrees to follow the contraceptive guidance in the protocol during the treatment period and for at least 6 weeks after the last dose of study vaccine
* Has a legally acceptable representative who understands the study procedures, alternate treatments available, and risks involved with the study and voluntarily agrees to participate by giving written informed consent/assent.

Exclusion Criteria:

* History of Invasive Pneumococcal Disease (positive blood culture, positive cerebrospinal fluid culture, or positive culture at another sterile site) or known history of other culture-positive pneumococcal disease within 3 years of Visit 1 (Day 1)
* Known hypersensitivity to any component of pneumococcal conjugate vaccine (PCV), or any diphtheria toxoid-containing vaccine
* Known or suspected impairment of immunological function
* History of congenital or acquired immunodeficiency
* Documented human immunodeficiency virus (HIV) infection
* History of autoimmune disease (including but not limited to systemic lupus erythematosus, antiphospholipid syndrome, Behcet's disease, autoimmune thyroid disease, polymyositis and dermatomyositis, scleroderma, or type 1 diabetes mellitus)
* Known coagulation disorder contraindicating intramuscular vaccination
* History of malignancy ≤5 years prior to signing informed consent/assent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* A WOCBP who has a positive urine or serum pregnancy test before the first vaccination at Visit 1 (Day 1)
* Received any PCV or pneumococcal polysaccharide vaccine <3 years before Visit 1 (Day 1)
* Five (5) years of age and has received <3 doses of PCV
* Receiving immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease. Note: hydroxyurea is permitted
* Received immunoglobulin within 6 months before receipt of study vaccine
* Participated in another clinical study of an investigational product within 2 months before the beginning or anytime during the duration of the current clinical study. Participants enrolled in observational studies may be included
* Recent history (within the last year) of more than 3 inpatient hospitalizations
* At the time of signing informed consent/assent, is a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence as assessed by the study investigator
* History or current evidence of any condition, therapy, lab abnormality or other circumstance that might expose the participant to risk by participating in the study, confound the results of the study, or interfere with the participant's participation for the full duration of the study in the opinion of the Investigator
* Is or has an immediate family member (eg, spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (19):
- United States (6):
  - Nemours/Alfred I. duPont Hospital for Children ( Site 0113), Wilmington, Delaware
  - Children's Healthcare of Atlanta ( Site 0100), Atlanta, Georgia
  - Children's Hospital of Michigan ( Site 0111), Detroit, Michigan
  - Newark Beth Israel Medical Center ( Site 0115), Newark, New Jersey
  - University of Rochester Medical Center ( Site 0105), Rochester, New York
  - Cincinnati Children's Hospital Medical Center ( Site 0101), Cincinnati, Ohio
- Brazil (3):
  - Santa Casa de Misericordia de Belo Horizonte ( Site 0200), Belo Horizonte, Minas Gerais
  - Hospital Santo Antonio - Obras Sociais Irma Dulce ( Site 0205), Salvador
  - Santa Casa de Misericordia de Sao Paulo ( Site 0202), São Paulo
- Colombia (2):
  - Clinica de la Costa Ltda. ( Site 0300), Barranquilla, Atlántico
  - Centro de Estudios en Infectologia Pediatrica SAS ( Site 0301), Cali, Valle del Cauca Department
- Dominican Republic (3):
  - Fundacion Dominicana de Perinatologia PRO BEBE INC ( Site 0402), Distrito Nacional, Santo Domingo Province
  - Clinical Research Republica Dominicana ( Site 0401), Santo Domingo
  - Caimed Dominicana S.A.S ( Site 0400), Santo Domingo
- Greece (2):
  - Agia Sophia Children s Hospital ( Site 0700), Athens
  - Hippokration General Hospital of Thessaloniki ( Site 0701), Thessaloniki
- Ospedale San Martino ( Site 0800), Genova, Italy
- Panama (2):
  - Cevaxin ( Site 0500), Panama City
  - Cevaxin ( Site 0502), Panama City

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Quinn CT, Wiedmann RT, Jarovsky D, Lopez-Medina E, Rodriguez HM, Papa M, Boggio G, Shou Q, Dagan R, Richmond P, Feemster K, McFetridge R, Tamms G, Lupinacci R, Musey L, Bickham K. Safety and immunogenicity of V114, a 15-valent pneumococcal conjugate vaccine, in children with SCD: a V114-023 (PNEU-SICKLE) study. Blood Adv. 2023 Feb 14;7(3):414-421. doi: 10.1182/bloodadvances.2022008037. PMID 36383730

RESULTS

PARTICIPANT FLOW:
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1.
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1.
Period: Overall Study
Arm/Group | V114 | Prevnar 13™
Started | 70 | 34
V114 or Prevnar 13™ Vaccination (Day 1) | 69 | 34
Completed | 65 | 34
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal By Parent/Guardian | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- V114: Participants received a single 0.5 mL IM injection of V114 on Day 1.
- Total: Total of all reporting groups
Arm/Group | V114 | Prevnar 13™ | Total
Number analyzed (Participants) | 70 | 34 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (3.5) | 10.8 (3.3) | 10.8 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 14 | 47
  Male | 37 | 20 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 24 | 68
  Not Hispanic or Latino | 26 | 10 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 3 | 12
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 25 | 63
  White | 10 | 2 | 12
  More than one race | 13 | 4 | 17
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited injection-site AEs included injection-site erythema (redness), injection-site induration (hard lump), injection-site pain (tenderness), and injection-site swelling.
Time Frame: Up to 14 days post-vaccination
Population: All randomized participants who received at least 1 dose of study vaccination
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 69 | 34
Percentage of participants
  Injection site erythema | 4.3 (0.9) [0.9 to 12.2] | 5.9 (0.7) [0.7 to 19.7]
  Injection site induration | 8.7 (3.3) [3.3 to 18.0] | 8.8 (1.9) [1.9 to 23.7]
  Injection site pain | 60.9 (48.4) [48.4 to 72.4] | 67.6 (49.5) [49.5 to 82.6]
  Injection site swelling | 27.5 (17.5) [17.5 to 39.6] | 35.3 (19.7) [19.7 to 53.5]

2. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited systemic AEs included arthralgia (joint pain), fatigue (tiredness), headache, myalgia (muscle pain), and urticaria (hives or welts).
Time Frame: Up to 14 days post-vaccination
Population: All randomized participants who received at least 1 dose of study vaccination
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 69 | 34
Percentage of participants
  Arthralgia | 2.9 (0.4) [0.4 to 10.1] | 8.8 (1.9) [1.9 to 23.7]
  Fatigue | 13.0 (6.1) [6.1 to 23.3] | 20.6 (8.7) [8.7 to 37.9]
  Headache | 24.6 (15.1) [15.1 to 36.5] | 17.6 (6.8) [6.8 to 34.5]
  Myalgia | 23.2 (13.9) [13.9 to 34.9] | 11.8 (3.3) [3.3 to 27.5]
  Urticaria | 0.0 (0.0) [0.0 to 5.2] | 2.9 (0.1) [0.1 to 15.3]

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event
Description: A serious adverse event (SAE) is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. SAEs that were reported by the investigator to be at least possibly related to the study vaccination were summarized.
Time Frame: Up to 6 months post-vaccination
Population: All randomized participants who received at least 1 dose of study vaccination
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 69 | 34
Percentage of participants | 0.0 (0.0) [0.0 to 5.2] | 0.0 (0.0) [0.0 to 10.3]

4. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Immunoglobulin G (IgG) at Day 30
Description: The GMC of IgG serotype-specific antibodies to the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™ and 2 serotypes (22F and 33F) unique to V114 were quantitated from participants' sera by a multiplex electrochemiluminescence (ECL) assay.
Time Frame: Day 30
Population: All randomized participants without deviations from the protocol that may have substantially affected the results of this immunogenicity endpoint and who had sufficient data to perform the analyses
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 69 | 34
μg/mL
  Serotype 1: number analyzed (Participants) | 66 | 32
  Serotype 1 | 2.12 [1.63 to 2.75] | 2.76 [1.95 to 3.91]
  Serotype 3: number analyzed (Participants) | 66 | 31
  Serotype 3 | 1.09 [0.87 to 1.38] | 1.07 [0.70 to 1.65]
  Serotype 4: number analyzed (Participants) | 66 | 31
  Serotype 4 | 1.58 [1.18 to 2.10] | 2.90 [2.00 to 4.20]
  Serotype 5: number analyzed (Participants) | 66 | 31
  Serotype 5 | 4.44 [3.19 to 6.17] | 6.56 [4.09 to 10.52]
  Serotype 6A: number analyzed (Participants) | 66 | 31
  Serotype 6A | 23.29 [17.22 to 31.52] | 15.97 [8.82 to 28.91]
  Serotype 6B: number analyzed (Participants) | 66 | 31
  Serotype 6B | 38.38 [28.53 to 51.64] | 22.94 [13.60 to 38.71]
  Serotype 7F: number analyzed (Participants) | 66 | 32
  Serotype 7F | 5.81 [4.42 to 7.64] | 4.65 [3.06 to 7.06]
  Serotype 9V: number analyzed (Participants) | 66 | 32
  Serotype 9V | 4.46 [3.44 to 5.78] | 5.36 [3.45 to 8.33]
  Serotype 14: number analyzed (Participants) | 66 | 31
  Serotype 14 | 16.03 [11.23 to 22.90] | 20.53 [12.39 to 34.03]
  Serotype 18C: number analyzed (Participants) | 66 | 32
  Serotype 18C | 6.11 [4.47 to 8.35] | 4.20 [2.66 to 6.62]
  Serotype 19A: number analyzed (Participants) | 66 | 32
  Serotype 19A | 19.86 [14.77 to 26.70] | 21.65 [14.45 to 32.44]
  Serotype 19F: number analyzed (Participants) | 66 | 32
  Serotype 19F | 13.88 [9.96 to 19.35] | 12.80 [9.10 to 18.01]
  Serotype 23F: number analyzed (Participants) | 63 | 31
  Serotype 23F | 5.38 [3.88 to 7.46] | 6.88 [4.01 to 11.83]
  Serotype 22F: number analyzed (Participants) | 66 | 30
  Serotype 22F | 7.30 [5.68 to 9.36] | 0.49 [0.33 to 0.73]
  Serotype 33F: number analyzed (Participants) | 66 | 32
  Serotype 33F | 4.46 [3.38 to 5.87] | 0.97 [0.62 to 1.51]

5. Secondary Outcome: Geometric Mean Titer (GMT) of Serotype-specific Opsonophagocytic Activity (OPA) at Day 30
Description: Sera from participants was used to measure GMT of 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™ and 2 serotypes (22F and 33F) unique to V114 using the multiplexed opsonophagocytic assay (MOPA).
Time Frame: Day 30
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dil
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 69 | 34
1/dil
  Serotype 1: number analyzed (Participants) | 51 | 22
  Serotype 1 | 484.0 [327.5 to 715.4] | 504.0 [254.8 to 997.0]
  Serotype 3: number analyzed (Participants) | 51 | 22
  Serotype 3 | 264.8 [193.4 to 362.4] | 234.3 [133.0 to 412.6]
  Serotype 4: number analyzed (Participants) | 51 | 22
  Serotype 4 | 4670.8 [2965.9 to 7355.6] | 7015.5 [3994.0 to 12322.6]
  Serotype 5: number analyzed (Participants) | 51 | 22
  Serotype 5 | 1383.9 [957.1 to 2000.9] | 1198.2 [638.1 to 2250.0]
  Serotype 6A: number analyzed (Participants) | 50 | 22
  Serotype 6A | 27305.7 [19797.6 to 37661.2] | 20277.1 [11740.2 to 35021.7]
  Serotype 6B: number analyzed (Participants) | 51 | 22
  Serotype 6B | 31560.4 [24134.1 to 41272.1] | 18531.0 [11024.7 to 31148.1]
  Serotype 7F: number analyzed (Participants) | 51 | 22
  Serotype 7F | 19411.5 [15195.9 to 24796.5] | 16928.1 [11107.4 to 25799.0]
  Serotype 9V: number analyzed (Participants) | 51 | 22
  Serotype 9V | 4561.8 [3240.7 to 6421.4] | 3941.7 [2659.6 to 5841.7]
  Serotype 14: number analyzed (Participants) | 51 | 22
  Serotype 14 | 6597.6 [4706.8 to 9248.0] | 8112.2 [4827.2 to 13632.8]
  Serotype 18C: number analyzed (Participants) | 50 | 22
  Serotype 18C | 9684.6 [6642.1 to 14120.7] | 5685.1 [3329.4 to 9707.6]
  Serotype 19A: number analyzed (Participants) | 51 | 22
  Serotype 19A | 14067.7 [9972.8 to 19843.9] | 9224.9 [5015.5 to 16967.1]
  Serotype 19F: number analyzed (Participants) | 51 | 22
  Serotype 19F | 4931.8 [3387.8 to 7179.7] | 3313.3 [2039.4 to 5383.1]
  Serotype 23F: number analyzed (Participants) | 50 | 22
  Serotype 23F | 17190.9 [12066.0 to 24492.4] | 19197.1 [10511.1 to 35061.1]
  Serotype 22F: number analyzed (Participants) | 51 | 19
  Serotype 22F | 7257.5 [5278.5 to 9978.3] | 1013.2 [477.4 to 2150.1]
  Serotype 33F: number analyzed (Participants) | 51 | 22
  Serotype 33F | 24013.6 [17612.4 to 32741.4] | 4824.8 [3216.3 to 7237.9]

6. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Serotype-specific IgG From Day 1 (Baseline) to Day 30
Description: IgG for the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™ and 2 serotypes unique to V114 (22F and 33F) was determined using an electrochemiluminescence assay. GMFR is defined as the geometric mean of the ratio of concentration at Day 30 after vaccination divided by concentration at baseline (Day 1, pre-vaccination).
Time Frame: Day 1 (Baseline) and Day 30
Population: All randomized participants without protocol deviations that could have substantially impacted the results of these immunogenicity analyses and who had sufficient data to perform the analyses
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 69 | 34
Ratio
  Serotype 1: number analyzed (Participants) | 66 | 30
  Serotype 1 | 6.2 [4.6 to 8.5] | 6.0 [3.7 to 9.9]
  Serotype 3: number analyzed (Participants) | 66 | 29
  Serotype 3 | 4.8 [3.5 to 6.6] | 4.1 [2.6 to 6.7]
  Serotype 4: number analyzed (Participants) | 66 | 29
  Serotype 4 | 6.0 [4.3 to 8.3] | 9.3 [5.4 to 16.2]
  Serotype 5: number analyzed (Participants) | 66 | 29
  Serotype 5 | 5.3 [3.8 to 7.4] | 6.4 [3.8 to 10.8]
  Serotype 6A: number analyzed (Participants) | 66 | 29
  Serotype 6A | 54.7 [37.9 to 78.9] | 40.6 [22.9 to 71.9]
  Serotype 6B: number analyzed (Participants) | 66 | 29
  Serotype 6B | 37.2 [25.8 to 53.6] | 25.0 [13.8 to 45.3]
  Serotype 7F: number analyzed (Participants) | 66 | 30
  Serotype 7F | 11.6 [8.3 to 16.0] | 9.8 [6.3 to 15.3]
  Serotype 9V: number analyzed (Participants) | 66 | 30
  Serotype 9V | 7.4 [5.3 to 10.3] | 8.1 [4.9 to 13.2]
  Serotype 14: number analyzed (Participants) | 65 | 29
  Serotype 14 | 10.8 [6.8 to 17.2] | 7.2 [3.5 to 14.8]
  Serotype 18C: number analyzed (Participants) | 66 | 30
  Serotype 18C | 10.8 [7.7 to 15.1] | 7.6 [4.5 to 12.8]
  Serotype 19A: number analyzed (Participants) | 66 | 30
  Serotype 19A | 8.2 [5.4 to 12.4] | 8.6 [5.0 to 14.9]
  Serotype 19F: number analyzed (Participants) | 66 | 30
  Serotype 19F | 8.3 [5.6 to 12.3] | 7.6 [4.5 to 12.8]
  Serotype 23F: number analyzed (Participants) | 63 | 29
  Serotype 23F | 9.3 [6.1 to 14.2] | 13.1 [7.4 to 23.4]
  Serotype 22F: number analyzed (Participants) | 66 | 28
  Serotype 22F | 15.0 [10.1 to 22.1] | 1.1 [0.9 to 1.3]
  Serotype 33F: number analyzed (Participants) | 66 | 30
  Serotype 33F | 9.0 [6.7 to 12.1] | 1.3 [1.0 to 1.7]

7. Secondary Outcome: GMFR in Serotype-specific OPA From Day 1 (Baseline) to Day 30
Description: Activity for the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™ and 2 serotypes unique to V114 (22F and 33F) was determined using a MOPA. GMFR is defined as the geometric mean of the ratio of concentration at Day 30 after vaccination divided by concentration at baseline (Day 1, pre-vaccination).
Time Frame: Day 1 (Baseline) and Day 30
Population: All randomized participants without protocol deviations that could have substantially affected the results of these immunogenicity analyses and who had sufficient data to perform the analyses
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- V114: Participants received a single 0.5 mL intramuscular IM injection of V114 on Day 1.
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 69 | 34
Ratio
  Serotype 1: number analyzed (Participants) | 49 | 20
  Serotype 1 | 24.1 [14.9 to 39.1] | 13.3 [5.1 to 34.2]
  Serotype 3: number analyzed (Participants) | 50 | 21
  Serotype 3 | 4.9 [3.5 to 7.0] | 3.1 [1.8 to 5.6]
  Serotype 4: number analyzed (Participants) | 49 | 21
  Serotype 4 | 10.2 [6.3 to 16.6] | 18.5 [8.8 to 38.9]
  Serotype 5: number analyzed (Participants) | 49 | 21
  Serotype 5 | 23.7 [15.0 to 37.5] | 13.8 [6.6 to 28.6]
  Serotype 6A: number analyzed (Participants) | 47 | 21
  Serotype 6A | 20.7 [13.3 to 32.1] | 11.2 [4.8 to 26.2]
  Serotype 6B: number analyzed (Participants) | 47 | 19
  Serotype 6B | 21.7 [12.7 to 36.9] | 13.7 [6.8 to 27.7]
  Serotype 7F: number analyzed (Participants) | 50 | 21
  Serotype 7F | 5.4 [3.8 to 7.7] | 5.4 [3.2 to 9.1]
  Serotype 9V: number analyzed (Participants) | 48 | 20
  Serotype 9V | 4.4 [3.0 to 6.5] | 6.1 [3.6 to 10.4]
  Serotype 14: number analyzed (Participants) | 50 | 21
  Serotype 14 | 6.9 [4.3 to 11.1] | 4.6 [2.1 to 10.2]
  Serotype 18C: number analyzed (Participants) | 45 | 20
  Serotype 18C | 14.0 [8.9 to 22.0] | 4.8 [2.5 to 9.3]
  Serotype 19A: number analyzed (Participants) | 50 | 21
  Serotype 19A | 9.0 [5.4 to 15.0] | 7.8 [4.4 to 14.0]
  Serotype 19F: number analyzed (Participants) | 50 | 20
  Serotype 19F | 6.4 [4.3 to 9.7] | 6.6 [3.3 to 12.9]
  Serotype 23F: number analyzed (Participants) | 48 | 20
  Serotype 23F | 10.4 [5.8 to 18.4] | 18.1 [8.8 to 37.1]
  Serotype 22F: number analyzed (Participants) | 48 | 17
  Serotype 22F | 6.5 [3.7 to 11.3] | 0.9 [0.7 to 1.2]
  Serotype 33F: number analyzed (Participants) | 50 | 21
  Serotype 33F | 3.8 [2.7 to 5.2] | 0.8 [0.7 to 1.0]

ADVERSE EVENTS:
Time Frame: Serious AEs and All-Cause Mortality: up to 6 months post-vaccination; Other AEs (non-serious): up to 14 days post-vaccination
Description: The safety analysis population included all randomized participants who received at least 1 dose of study vaccination.
  The analysis population for All-Cause Mortality included all randomized participants.
Groups:
- Prevnar 13: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1.
Arm/Group | V114 | Prevnar 13
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/34
Serious Adverse Events (participants affected / at risk) | 13/69 | 8/34
Other Adverse Events (participants affected / at risk) | 52/69 | 27/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=69) | Prevnar 13 (N=34)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 7 (9) | 6 (7)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medical observation (Investigations) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=69) | Prevnar 13 (N=34)
Fatigue (General disorders) | 9 (9) | 7 (7)
Injection site erythema (General disorders) | 3 (3) | 2 (2)
Injection site induration (General disorders) | 6 (6) | 3 (3)
Injection site pain (General disorders) | 42 (48) | 23 (25)
Injection site swelling (General disorders) | 19 (21) | 12 (14)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 16 (20) | 4 (7)
Headache (Nervous system disorders) | 17 (25) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT03731182/Prot_SAP_000.pdf